CLINICAL TRIAL: NCT01337986
Title: Dalfampridine After Optic Neuritis to Improve Visual Function in Multiple Sclerosis
Brief Title: Ampyra for Optic Neuritis in Multiple Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Ampyra Vision 2011 RTN; WU HRPO# : 201104126 (Other: Washington University HRPO)
Record Dates: First submitted 2011-04-13; First posted 2011-04-19 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis; Optic Neuritis
Keywords: Multiple Sclerosis; Optic Neuritis; Ampyra; Dalfampridine; Fampridine; Remote Optic Neuritis; Contrast Sensitivity; Treatment
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group B: Dalfampridine First (Active Comparator): Dalfampridine/Placebo: Weeks 1-3: Dalfampridine 10mg (1 tablet) every 12 hours for 3 weeks. Weeks 4-5: 2 weeks of wash-out. Weeks 5-8: Placebo (sugar pill) 1 tablet every 12 hours for 3 weeks.
  Interventions: Drug: Dalfampridine/Placebo
- Group A: Dalfampridine Second (Active Comparator): Placebo/Dalfampridine: Weeks 1-3: Placebo (sugar pill) 1 tablet every 12 hours for 3 weeks. Weeks 4-5: 2 weeks of wash-out. Weeks 6-8: Dalfampridine 10mg (1 tablet) every 12 hours for 3 weeks
  Interventions: Drug: Placebo/Dalfampridine

INTERVENTIONS:
Drug: Dalfampridine/Placebo — Weeks 1-3: Dalfampridine 10mg (1 tablet) every 12 hours for 3 weeks. Weeks 4-5: 2 weeks of wash-out. Weeks 5-8: Placebo (sugar pill) 1 tablet every 12 hours for 3 weeks.
  Other Names: Ampyra (R); Fampridine
  Arms: Group B: Dalfampridine First
Drug: Placebo/Dalfampridine — Weeks 1-3: Placebo (sugar pill) 1 tablet every 12 hours for 3 weeks. Weeks 4-5: 2 weeks of wash-out. Weeks 6-8: Dalfampridine 10mg (1 tablet) every 12 hours for 3 weeks.
  Other Names: Ampyra (R); Fampridine
  Arms: Group A: Dalfampridine Second

SUMMARY:
Fifty subjects will be enrolled in this Phase II, investigator-initiated, randomized and blinded cross-over trial of dalfampridine of 8 weeks duration The study will test the hypothesis that dalfampridine, when administered to subjects with incomplete visual recovery after optic neuritis from MS, will result in symptomatic improvement in visual function. The study will consist of one screening/baseline visit, one visit during treatment with active drug, and one visit on placebo. After the baseline visit, subjects will be randomly assigned to receive study medication or placebo for the first three weeks, followed by a two week wash-out, and then treatment reallocation for the latter three weeks.

DETAILED DESCRIPTION:
Optic neuritis (ON) is the presenting feature of multiple sclerosis (MS) in 15% of cases, and occurs over the disease course in 50% of patients.1-3 Vision remains a major concern for MS patients, as visual dysfunction leads to lower quality of life.4-6 Despite the high prevalence of ON in MS, treatment and management options remain limited. Although intravenous glucocorticoids are employed to aid recovery of an acute episode of ON, no convincing evidence supports their efficacy in altering the degree of long-term recovery.7 Although some individuals with ON can have a dramatic recovery from blindness, ON often impairs visual function permanently. In the Optic Neuritis Treatment Trial, 63% reported that vision had not returned to normal after 6 months, and 20% had vision worse than 20/20 after 5 years of follow-up.8, 9 Visual impairment creates difficulties at home and work, leading to decreased independence and impaired mobility within the community. Visual dysfunction in combination with MS impairments within cerebellar and proprioceptive systems can be particularly disabling.

Optic neuritis classically impairs one's ability to read print or a computer screen, to drive in bright or low light, and to appreciate colors and contrasts. Unfortunately, when optic neuritis results in lasting impairment, there are no pharmacologic therapies to restore vision. Low vision specialists may provide magnifying glasses, brighter lights, and advice to optimize the position of objects at home and in the workplace. Better treatment options are needed to improve visual function.

Ampyra (dalfampridine) is a potassium-channel antagonist, with a mechanism-of-action to improve nerve conduction in demyelinated axons, resulting in an electrophysiologic and clinical benefit.10-22 Demyelinated axons within the anterior visual pathway would be a prime and ideal target to study the effects of Ampyra. In fact, Stefoski et al demonstrated visual function benefit in an open-label study of IV 4-aminopyridine in 12 subjects.21 The optic nerves are a well-defined white-matter tract, commonly affected in MS, and with clear clinical outcome measures. In addition, visual evoked potentials (VEPs) can be included within the study design as a secondary endpoint, to confirm improved nerve conduction. Because VEPs are such a precise, reliable, and accepted measure of demyelination, the anterior visual pathway is the ideal in vivo human system to study the electro-physiologic effects of a therapeutic such as Ampyra.

Hypothesis 1: Dalfampridine treatment will improve visual function, measured by the 5% ETDRS contrast sensitivity chart, in subjects with long-term visual impairment secondary to optic neuritis from MS.

Hypothesis 2: Dalfampridine treatment will reduce visual evoked potential P100 latency following remote optic neuritis.

Hypothesis 3: Dalfampridine treatment will result in an improvement in secondary endpoints, including visual fields, high contrast visual acuity, color vision, and quality of life.

The study will be conducted at the Department of Neurology and Neurosurgery, Washington University School of Medicine, St. Louis, the institution at which Dr. Naismith is based. The MS patients will come from the 1800 active MS patients in our clinic and the 3500 in the St. Louis area.

Fifty subjects will be enrolled in this Phase II, investigator-initiated, randomized and blinded cross-over trial of dalfampridine of 8 weeks duration (Table 1). The study will test the hypothesis that dalfampridine, when administered to subjects with incomplete visual recovery after optic neuritis from MS, will result in symptomatic improvement in visual function. The study will consist of one screening/baseline visit, one visit during treatment with active drug, and one visit on placebo. After the baseline visit, subjects will be randomly assigned to receive study medication or placebo for the first three weeks, followed by a two week wash-out, and then treatment reallocation for the latter three weeks.

ELIGIBILITY:
Inclusion criteria are:

1. At least one previous clinical episode of optic neuritis,
2. the last episode of ON must have occurred at least 12 months prior to study entry,
3. clinically definite MS, defined by the revised McDonald criteria, 23
4. ages 18-70,
5. visual acuity greater than or equal to 20/30
6. must be able to read at least 2 of the 5 letters on the top line of the 5% ETDRS chart (logMAR 0.96) at 3 meters, 2 meters or 1 meter, and
7. must have sufficient cognitive function to understand the consent process and to reliably perform all clinical assessments

Exclusion criteria are:

1. Any ophthalmologic condition, other than ON, which can affect vision, including nystagmus in primary position of gaze,
2. history of seizures or spells with altered level of consciousness,
3. pregnancy or breast feeding,
4. an MS exacerbation or use of glucocorticoids within 3 months of entry,
5. a history of moderate to severe renal insufficiency,
6. previous use of 4-aminopyridine, in any formulation, in the prior 4 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Naismith, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University (John L. Trotter MS Center), St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frohman EM, Frohman TC, Zee DS, McColl R, Galetta S. The neuro-ophthalmology of multiple sclerosis. Lancet Neurol. 2005 Feb;4(2):111-21. doi: 10.1016/S1474-4422(05)00992-0. PMID 15664543
- [Background] Arnold AC. Evolving management of optic neuritis and multiple sclerosis. Am J Ophthalmol. 2005 Jun;139(6):1101-8. doi: 10.1016/j.ajo.2005.01.031. PMID 15953446
- [Background] Balcer LJ. Clinical practice. Optic neuritis. N Engl J Med. 2006 Mar 23;354(12):1273-80. doi: 10.1056/NEJMcp053247. No abstract available. PMID 16554529
- [Background] Ma SL, Shea JA, Galetta SL, Jacobs DA, Markowitz CE, Maguire MG, Balcer LJ. Self-reported visual dysfunction in multiple sclerosis: new data from the VFQ-25 and development of an MS-specific vision questionnaire. Am J Ophthalmol. 2002 May;133(5):686-92. doi: 10.1016/s0002-9394(02)01337-5. PMID 11992867
- [Background] Noble J, Forooghian F, Sproule M, Westall C, O'Connor P. Utility of the National Eye Institute VFQ-25 questionnaire in a heterogeneous group of multiple sclerosis patients. Am J Ophthalmol. 2006 Sep;142(3):464-8. doi: 10.1016/j.ajo.2006.04.051. PMID 16935592
- [Background] Mowry EM, Loguidice MJ, Daniels AB, Jacobs DA, Markowitz CE, Galetta SL, Nano-Schiavi ML, Cutter GR, Maguire MG, Balcer LJ. Vision related quality of life in multiple sclerosis: correlation with new measures of low and high contrast letter acuity. J Neurol Neurosurg Psychiatry. 2009 Jul;80(7):767-72. doi: 10.1136/jnnp.2008.165449. Epub 2009 Feb 23. PMID 19240050
- [Background] Beck RW, Cleary PA, Anderson MM Jr, Keltner JL, Shults WT, Kaufman DI, Buckley EG, Corbett JJ, Kupersmith MJ, Miller NR, et al. A randomized, controlled trial of corticosteroids in the treatment of acute optic neuritis. The Optic Neuritis Study Group. N Engl J Med. 1992 Feb 27;326(9):581-8. doi: 10.1056/NEJM199202273260901. PMID 1734247
- [Background] Visual function 5 years after optic neuritis: experience of the Optic Neuritis Treatment Trial. The Optic Neuritis Study Group. Arch Ophthalmol. 1997 Dec;115(12):1545-52. PMID 9400788
- [Background] Cleary PA, Beck RW, Bourque LB, Backlund JC, Miskala PH. Visual symptoms after optic neuritis. Results from the Optic Neuritis Treatment Trial. J Neuroophthalmol. 1997 Mar;17(1):18-23; quiz 24-8. doi: 10.1016/s0002-9394(14)70814-1. PMID 9093956
- [Background] Goodman AD, Brown TR, Krupp LB, Schapiro RT, Schwid SR, Cohen R, Marinucci LN, Blight AR; Fampridine MS-F203 Investigators. Sustained-release oral fampridine in multiple sclerosis: a randomised, double-blind, controlled trial. Lancet. 2009 Feb 28;373(9665):732-8. doi: 10.1016/S0140-6736(09)60442-6. PMID 19249634
- [Background] Fujihara K, Miyoshi T. The effects of 4-aminopyridine on motor evoked potentials in multiple sclerosis. J Neurol Sci. 1998 Jul 15;159(1):102-6. doi: 10.1016/s0022-510x(98)00143-9. PMID 9700711
- [Background] Schwid SR, Petrie MD, McDermott MP, Tierney DS, Mason DH, Goodman AD. Quantitative assessment of sustained-release 4-aminopyridine for symptomatic treatment of multiple sclerosis. Neurology. 1997 Apr;48(4):817-21. doi: 10.1212/wnl.48.4.817. PMID 9109861
- [Background] Davis FA, Stefoski D, Quandt FN. Mechanism of action of 4-aminopyridine in the symptomatic treatment of multiple sclerosis. Ann Neurol. 1995 May;37(5):684. doi: 10.1002/ana.410370524. No abstract available. PMID 7755367
- [Background] Bever CT Jr, Young D, Anderson PA, Krumholz A, Conway K, Leslie J, Eddington N, Plaisance KI, Panitch HS, Dhib-Jalbut S, et al. The effects of 4-aminopyridine in multiple sclerosis patients: results of a randomized, placebo-controlled, double-blind, concentration-controlled, crossover trial. Neurology. 1994 Jun;44(6):1054-9. doi: 10.1212/wnl.44.6.1054. PMID 8208399
- [Background] Polman CH, Bertelsmann FW, van Loenen AC, Koetsier JC. 4-aminopyridine in the treatment of patients with multiple sclerosis. Long-term efficacy and safety. Arch Neurol. 1994 Mar;51(3):292-6. doi: 10.1001/archneur.1994.00540150090022. PMID 8129642
- [Background] van Diemen HA, Polman CH, van Dongen MM, Nauta JJ, Strijers RL, van Loenen AC, Bertelsmann FW, Koetsier JC. 4-Aminopyridine induces functional improvement in multiple sclerosis patients: a neurophysiological study. J Neurol Sci. 1993 Jun;116(2):220-6. doi: 10.1016/0022-510x(93)90329-w. PMID 8336169
- [Background] van Diemen HA, Polman CH, van Dongen TM, van Loenen AC, Nauta JJ, Taphoorn MJ, van Walbeek HK, Koetsier JC. The effect of 4-aminopyridine on clinical signs in multiple sclerosis: a randomized, placebo-controlled, double-blind, cross-over study. Ann Neurol. 1992 Aug;32(2):123-30. doi: 10.1002/ana.410320203. PMID 1510353
- [Background] Stefoski D, Davis FA, Fitzsimmons WE, Luskin SS, Rush J, Parkhurst GW. 4-Aminopyridine in multiple sclerosis: prolonged administration. Neurology. 1991 Sep;41(9):1344-8. doi: 10.1212/wnl.41.9.1344. PMID 1891078
- [Background] Polman CH, van Diemen HA, van Dongen MM, Koetsier JC, van Loenen AC, van Walbeek HK. 4-Aminopyridine in multiple sclerosis. Ann Neurol. 1990 Oct;28(4):589. doi: 10.1002/ana.410280421. No abstract available. PMID 2082971
- [Background] Davis FA, Stefoski D, Rush J. Orally administered 4-aminopyridine improves clinical signs in multiple sclerosis. Ann Neurol. 1990 Feb;27(2):186-92. doi: 10.1002/ana.410270215. PMID 2317014
- [Background] Polman CH, Reingold SC, Edan G, Filippi M, Hartung HP, Kappos L, Lublin FD, Metz LM, McFarland HF, O'Connor PW, Sandberg-Wollheim M, Thompson AJ, Weinshenker BG, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2005 revisions to the "McDonald Criteria". Ann Neurol. 2005 Dec;58(6):840-6. doi: 10.1002/ana.20703. PMID 16283615
- [Background] Jones RE, Heron JR, Foster DH, Snelgar RS, Mason RJ. Effects of 4-aminopyridine in patients with multiple sclerosis. J Neurol Sci. 1983 Aug-Sep;60(3):353-62. doi: 10.1016/0022-510x(83)90145-4. PMID 6631441
- [Background] Vollmer T, Henney HR 3rd. Pharmacokinetics and tolerability of single escalating doses of fampridine sustained-release tablets in patients with multiple sclerosis: a Phase I-II, open-label trial. Clin Ther. 2009 Oct;31(10):2206-14. doi: 10.1016/j.clinthera.2009.10.008. PMID 19922891
- [Background] Vollmer T, Blight AR, Henney HR 3rd. Steady-state pharmacokinetics and tolerability of orally administered fampridine sustained-release 10-mg tablets in patients with multiple sclerosis: a 2-week, open-label, follow-up study. Clin Ther. 2009 Oct;31(10):2215-23. doi: 10.1016/j.clinthera.2009.10.007. PMID 19922892
- [Background] Beck RW, Ruchman MC, Savino PJ, Schatz NJ. Contrast sensitivity measurements in acute and resolved optic neuritis. Br J Ophthalmol. 1984 Oct;68(10):756-9. doi: 10.1136/bjo.68.10.756. PMID 6477856
- [Background] Trobe JD, Beck RW, Moke PS, Cleary PA. Contrast sensitivity and other vision tests in the optic neuritis treatment trial. Am J Ophthalmol. 1996 May;121(5):547-53. doi: 10.1016/s0002-9394(14)75429-7. PMID 8610798
- [Background] Farnsworth D. The Farnsworth-Munsell 100-hue and dichotomous tests for color vision. J Opt Soc Am 1943;33:568-574.
- [Background] Naismith RT, Tutlam NT, Xu J, Klawiter EC, Shepherd J, Trinkaus K, Song SK, Cross AH. Optical coherence tomography differs in neuromyelitis optica compared with multiple sclerosis. Neurology. 2009 Mar 24;72(12):1077-82. doi: 10.1212/01.wnl.0000345042.53843.d5. PMID 19307541
- [Background] Naismith RT, Tutlam NT, Xu J, Shepherd JB, Klawiter EC, Song SK, Cross AH. Optical coherence tomography is less sensitive than visual evoked potentials in optic neuritis. Neurology. 2009 Jul 7;73(1):46-52. doi: 10.1212/WNL.0b013e3181aaea32. PMID 19564583
- [Background] Naismith RT, Xu J, Tutlam NT, Trinkaus K, Cross AH, Song SK. Radial diffusivity in remote optic neuritis discriminates visual outcomes. Neurology. 2010 May 25;74(21):1702-10. doi: 10.1212/WNL.0b013e3181e0434d. PMID 20498438
- [Background] Naismith RT, Xu J, Tutlam NT, Scully PT, Trinkaus K, Snyder AZ, Song SK, Cross AH. Increased diffusivity in acute multiple sclerosis lesions predicts risk of black hole. Neurology. 2010 May 25;74(21):1694-701. doi: 10.1212/WNL.0b013e3181e042c4. PMID 20498437
- [Background] Naismith RT, Xu J, Tutlam NT, Snyder A, Benzinger T, Shimony J, Shepherd J, Trinkaus K, Cross AH, Song SK. Disability in optic neuritis correlates with diffusion tensor-derived directional diffusivities. Neurology. 2009 Feb 17;72(7):589-94. doi: 10.1212/01.wnl.0000335766.22758.cd. Epub 2008 Dec 10. PMID 19073948
- [Background] Naismith RT, Shepherd JB, Weihl CC, Tutlam NT, Cross AH. Acute and bilateral blindness due to optic neuropathy associated with copper deficiency. Arch Neurol. 2009 Aug;66(8):1025-7. doi: 10.1001/archneurol.2009.70. PMID 19667226
- [Background] Vanden Bosch ME, Wall M. Visual acuity scored by the letter-by-letter or probit methods has lower retest variability than the line assignment method. Eye (Lond). 1997;11 ( Pt 3):411-7. doi: 10.1038/eye.1997.87. PMID 9373488
- [Background] Acorda Therapeutics. AMPRYA package insert (2010).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the John L Trotter Multiple Sclerosis (MS) Clinic at Washington University and through email blasts from the Gateway (St. Louis) MS Chapter. 53 participants meet the pre-screening criteria and signed an informed consent to be screened for the study.
Pre-assignment Details: Patients whose vision did not meet study criteria at the first visit in the affected eye or who had had steroids within 3 months of study entry were considered screen failures (n =7).Treatment group was randomly assigned by the pharmacist using a randomization table generated by a probability model.
Groups:
- Group B: Dalfampridine/Placebo: Dalfampridine/Placebo: Weeks 1-3: Dalfampridine 10mg (1 tablet) every 12 hours for 3 weeks. Weeks 4-5: 2 weeks of wash-out. Weeks 5-8: Placebo (sugar pill) 1 tablet every 12 hours for 3 weeks.
- Group A: Placebo/Dalfampridine: Placebo/Dalfampridine: Weeks 1-3: Placebo (sugar pill) 1 tablet every 12 hours for 3 weeks. Weeks 4-5: 2 weeks of wash-out. Weeks 6-8: Dalfampridine 10mg (1 tablet) every 12 hours for 3 weeks.
Period: Overall Study
Arm/Group | Group B: Dalfampridine/Placebo | Group A: Placebo/Dalfampridine
Started | 23 | 23
Completed | 20 | 18
Not Completed | 3 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Population: All patients that were randomized and included in the per-protocol analysis (compliantly completed 3 visits on assigned treatment).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group B: Dalfampridine/Placebo | Group A: Placebo/Dalfampridine | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (10.7) | 50.7 (10.2) | 47.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 16 | 13 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38
MS Subtype [Number; unit: participants]
  Relapsing Remitting MS (RRMS) | 17 | 15 | 32
  Secondary Progressive MS (SPMS) | 3 | 3 | 6
Clinical Episodes of ON [Median (Full Range); unit: Number of episodes] | 1 [1 to 4] | 1 [1 to 4] | 1 [1 to 4]
Baseline 5% Sloan Chart [Median (Full Range); unit: Number of Letters] | 22 [2 to 46] | 20 [2 to 45] | 21 [2 to 46]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Dalfampridine on Visual Function by Early Diabetic Treatment Retinopathy Study (EDTRS) 5% Contrast Sensitivity Scores
Description: Per Protocol Analysis to assess differences in EDTRS 5% Contrast Sensitivity (LogMAR) Scores at visits 2 and 3 Relative to Visit 1 on patients taking Dalfampridine vs Placebo.
Time Frame: Visit 1 (Week 0), Visit 2 (Week 3) and Visit 3 (Week 8)
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: LogMAR Score
Units Other Than Participants: eligible eyes
Groups:
- Group B: Dalfampridine; Group B: Placebo: Dalfampridine/Placebo: Weeks 1-3: Dalfampridine 10mg (1 tablet) every 12 hours for 3 weeks. Weeks 4-5: 2 weeks of wash-out. Weeks 5-8: Placebo (sugar pill) 1 tablet every 12 hours for 3 weeks.
- Group A: Placebo; Group A: Dalfampridine: Placebo/Dalfampridine: Weeks 1-3: Placebo (sugar pill) 1 tablet every 12 hours for 3 weeks. Weeks 4-5: 2 weeks of wash-out. Weeks 6-8: Dalfampridine 10mg (1 tablet) every 12 hours for 3 weeks.
Arm/Group | Group B: Dalfampridine | Group B: Placebo | Group A: Placebo | Group A: Dalfampridine
Number analyzed (Participants) | 20 | 20 | 18 | 18
Number analyzed (eligible eyes) | 30 | 30 | 29 | 29
LogMAR Score | -0.04 (0.02) | -0.06 (0.02) | -0.08 (0.02) | -0.06 (0.02)
Statistical Analysis 1: Comparison: Group B: Dalfampridine vs Group B: Placebo vs Group A: Placebo vs Group A: Dalfampridine; Per protocol Analysis; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis
Statistical Analysis 2: Comparison: Group B: Dalfampridine vs Group B: Placebo vs Group A: Placebo vs Group A: Dalfampridine; Change in EDTRS between Visits 2 and 3; Test type: Superiority or Other; p = .29, Mixed Models Analysis

2. Primary Outcome: Efficacy of Dalfampridine on Visual Function Assessed by Change From Baseline in Raw Letters by EDTRS 5% Contrast Sensitivity
Description: Per Protocol Analysis to assess difference in number of letters on the EDTRS 5% Contrast Sensitivity (LogMAR) Chart scores at visits 2 and 3 Relative to Visit 1
Time Frame: Visit 1 (Week 0), Visit 2 (Week 3) and Visit 3 (Week 8)
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eligible eyes
Arm/Group | Group B: Dalfampridine | Group B: Placebo | Group A: Placebo | Group A: Dalfampridine
Number analyzed (Participants) | 20 | 20 | 18 | 18
Number analyzed (eligible eyes) | 30 | 30 | 29 | 29
letters | 2 (1) | 2 (1) | 4 (1) | 3 (1)

3. Primary Outcome: Difference in EDTRS 5% Contrast Sensitivity (LogMAR Score) at Visits 2 and 3 Relative to Visit 1
Description: Intent to treat analysis of treatment effect in primary endpoint EDTRS 5% Contrast Sensitivity. Improvement from baseline scores.
Time Frame: Visit 1 (Week 0), Visit 2 (Week 3) and Visit 3 (Week 8)
Population: Intent To Treat Population, scores from morning and afternoon were averaged.
Measure: Mean (Standard Deviation); unit: 5% Contrast LogMAR Score
Groups:
- Dalfampridine; Placebo: Patient Assessments while on Dalfampridine
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 46 | 46
5% Contrast LogMAR Score | 0.06 (0.02) | 0.05 (0.02)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Null hypothesis: there will be no difference in the change relevant to baseline (visit 1) in EDTRS 5% contrast sensitivity with dalfampridine vs placebo; Test type: Superiority or Other; p = .64, Mixed Models Analysis; Mean Difference (Final Values) = 0.008, Standard Error of Mean 0.01
Statistical Analysis 2: Comparison: Dalfampridine vs Placebo; Null hypothesis for period effect: there will be no difference in the change relevant to baseline (visit 1) in EDTRS 5% contrast sensitivity for those who started on dalfampridine and crossed over to placebo, compared to those who started on placebo and crossed over to dalfampridine; Test type: Superiority or Other; p = 0.11, Mixed Models Analysis

4. Secondary Outcome: Percentage of Eyes That Improved by 2 Lines (10 Letters) on the Sloan 5% Contrast Sensitivity Chart
Time Frame: Visit 1 (Week 0), Visit 2 (Week 3) and Visit 3 (Week 8)
Measure: Number (95% Confidence Interval); unit: Percentages of eyes that improved
Units Other Than Participants: Number of Eyes
Groups:
- Dalfampridine: Improvement while on Dalfampridine (not placebo)
- Placebo: Improvement while on Placebo (not dalfampridine)
- Both: Improvement when taking Dalfampridine or Placebo (improvement with any treatment)
- None: No Improvement on Dalfampridine/Placebo.
Arm/Group | Dalfampridine | Placebo | Both | None
Number analyzed (Participants) | 46 | 46 | 46 | 46
Number analyzed (Number of Eyes) | 72 | 72 | 72 | 72
Percentages of eyes that improved | 9.7 [4.0 to 19.0] | 11.1 [4.9 to 20.7] | 11.1 [4.9 to 20.7] | 68.1 [56.0 to 78.6]
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo vs Both vs None; Test type: Superiority or Other; p = 0.93, Regression, Logistic

5. Secondary Outcome: Percentage of Eyes That Improved by One-line (5 Letters)
Description: Percentage of eyes that improved by one-line (5 letters) on the 5% contrast sensitivity chart
Time Frame: Visit 1 (Week 0), Visit 2 (Week 3) and Visit 3 (Week 8)
Population: Proportion as the Percent of Eyes Improved by 1 Line
Measure: Number (95% Confidence Interval); unit: Percent of Eyes
Units Other Than Participants: Number of Eyes
Groups:
- Dalfampridine: Improvement while on Dalfampridine
- Placebo: Improvement while on Placebo
- Both: Improvement on Dalfampridine and Placebo
- Neither: No Improvement on Dalfampridine or Placebo
Arm/Group | Dalfampridine | Placebo | Both | Neither
Number analyzed (Participants) | 38 | 38 | 38 | 38
Number analyzed (Number of Eyes) | 72 | 72 | 72 | 72
Percent of Eyes | 11.1 [4.9 to 20.7] | 15.3 [7.9 to 25.7] | 37.5 [26.4 to 49.7] | 36.1 [25.1 to 48.3]
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo vs Both; Test type: Superiority or Other; p = .34, Regression, Logistic

6. Secondary Outcome: Visual Evoked Potential P100 Latency Per Treatment Arm
Description: Visual evoked potential 60min P100 latency on dalfampridine vs. placebo.
Time Frame: Visit 1 (Week 0), Visit 2 (Week 3) and Visit 3 (Week 8)
Population: per protocol
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 38 | 38
milliseconds | 121.6 (2.4) | 120.2 (2.4)

7. Secondary Outcome: Odds Ratio Quartile of Visual Field Index
Description: The Visual Field Index (VFI) is a global index that assigns a number between 1% to 100% based on an aggregate percentage of visual function, with 100% being a perfect age-adjusted visual field.
  Probability of falling in the best quartile for visual field (VFI) measures (Q1), relative to the three next quartiles for worse VFIs (Q2-4), while on Dalfampridine vs Placebo. Due to the clustered observations at different times in a cross-over design, the visual field data is not suited to a normal theory model and should not be expressed as a continuous variable. Thus, a categorical model that uses a multinomial distribution for measurement of 4 categories was selected for proper statistical modeling, with results expressed as odds ratios.
Time Frame: Visit 1 (Week 0 - baseline), Visit 2 (Week 3 - post intervention 1) and Visit 3 (Week 8 - post intervention 2)
Measure: Mean (Standard Deviation); unit: Visual Field Index % of normal vision
Units Other Than Participants: eligible eyes
Groups:
- Dalfampridine Then Placebo: Weeks 1-3 Dalfampridine 10 mg Twice Daily, Weeks 6-8 Placebo Twice Daily
- Placebo Then Dalfampridine: Weeks 1-3 Placebo Twice Daily, Weeks 6-8 Dalfampridine 10 mg Twice Daily
Arm/Group | Dalfampridine Then Placebo | Placebo Then Dalfampridine
Number analyzed (Participants) | 20 | 18
Number analyzed (eligible eyes) | 30 | 29
Visual Field Index % of normal vision
  Baseline (Visit 1) | 77.53 (29.84) | 85.38 (86.65)
  Post Intervention 1 (Visit 2) | 78.50 (28.30) | 86.65 (22.64)
  Post Intervention 2 (Visit 3) | 79.71 (28.57) | 86.00 (22.75)
Statistical Analysis 1: Comparison: Dalfampridine Then Placebo vs Placebo Then Dalfampridine; Test type: Superiority or Other; p = 0.04, Regression, Logistic — Probability of being in the lowest quartile for Visual Field Index deficits; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.02 to 2.10] — Odds Ratio for Visual Field Index

8. Secondary Outcome: Changes in Color Vision Total Error Score From Baseline Based Upon the Farnsworth Munsell Hue 100 Sort Test (FM100).
Description: Dalfampridine will change color vision Total Error Scores from baseline on the Farnsworth Munsell 100 Hue Sort Test. Farnsworth Munsell 100 Hue Test requires placing 100 color palettes in the correct order based upon color hue. Scores are determined by the frequency and severity of any displacement in the correct order. One error equates to one misplaced hue, by one step or position. An error score greater than 500 indicates virtually no color discrimination. An error score of 0 indicates no errors in ordering the hues. A Total Error Score of 0 to 128 could be seen in a normal population.
Time Frame: Visit 1 (Week 0 - baseline), Visit 2 (Week 3 - postintervention 1) and Visit 3 (Week 8 - post intervention 2)
Population: per protocol
Measure: Mean (Full Range); unit: FM100 Total Error Score
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 38 | 38
FM100 Total Error Score | -13.0 [-15.0 to -11.0] | -10.6 [-28.3 to -7.1]
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Test type: Superiority or Other; p = 0.94, Regression, Logistic

9. Secondary Outcome: Dalfampridine Effect on Quality of Life Change From Baseline.
Description: Dalfampridine treatment will result in change in quality of life. The National Eye Institute Visual Function Questionnaire consists of 25 questions characterizing visual function at home and in the community. Score ranges from 100 (best) to 0 (worst).
Time Frame: Visit 1 (Week 0), Visit 2 (Week 3) and Visit 3 (Week 8)
Measure: Median (Full Range); unit: NEI VFQ percentage
Groups:
- Dalfampridine: Study participants on dalfampridine
- Placebo: Study participants on placebo
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 38 | 38
NEI VFQ percentage | 0 [-40.0 to 30.0] | 0 [-35.0 to 302.5]
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Difference in Pelli- Robson Score at Visits 2 and 3 Relative to Visit 1
Description: Difference in Pelli- Robson Score at Visits 2 and 3 Relative to Visit 1 on Dalfampridine vs Placebo. Pelli-Robson is scored based upon the numbers read on the chart converted to LogMAR units. The scale is 0.00 (worst) to 2.35 (best).
Time Frame: Visit 1 (Week 0), Visit 2 (Week 3) and Visit 3 (Week 8)
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Number of Eyes
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 38 | 38
Number analyzed (Number of Eyes) | 60 | 60
units on a scale | 0.07 (0.02) | 0.06 (0.02)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Test type: Superiority or Other; p = 0.72, Regression, Linear

11. Primary Outcome: Change From Baseline in Raw Letters by EDTRS 5% Contrast Sensitivity
Description: Intent to treat analysis of treatment effect in primary endpoint EDTRS 5% Contrast Sensitivity. Change in the number of letters able to read while on Dalfampridine and Placebo relative to their baseline scores.
Time Frame: Visit 1 (Week 0), Visit 2 (Week 3) and Visit 3 (Week 8)
Population: Intent To Treat Population, scores from morning and afternoon were averaged.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 46 | 46
letters | 3 (1) | 2.5 (1)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Only unexpected and and reasonably related events were recorded. Adverse events related to known side effects of dalfampridine (listed in the package insert) or the patients prior medical history are not recorded. There were no events that warranted modification to the consent for the duration of the study. All adverse events (four) occurred while taking dalfmapridine during this cross-over study.
Groups:
- Dalfampridine: Participants assigned to received dalfampridine.
- Placebo: Participants assigned to received placebo.
Arm/Group | Dalfampridine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 4/46 | 0/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalfampridine (N=46) | Placebo (N=46)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Pilot study with relatively small number of patients compared to a phase III study. Cross-over design may be inferior to placebo-controlled parallel cohort study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days